CLINICAL TRIAL: NCT05255510
Title: Reducing Risk of Acute Kidney Injury After Living Donor Hepatectomy by Protocolized Fluid Restriction: Single-center Experience
Brief Title: Risk of Acute Kidney Injury in Living Liver Donor Surgery
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Collaborators: Elvan Onur Kırımker (Unknown); Sevcan Büyük (Unknown); Elif Beyza Baskan (Unknown); Ali Abbas Yılmaz (Unknown); Deniz Balcı (Unknown); Kaan Karayalçın (Unknown); Mustafa Kemal Bayar (Unknown)
Responsible Party: Principal Investigator, Süheyla Karadağ Erkoç, Anesthesiology and Reanimation, Ankara University
Other Study IDs: AnkaraUni
Record Dates: First submitted 2022-02-14; First posted 2022-02-24 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Acute Kidney Injury; Liver Transplant; Complications; Fluid and Electrolyte Imbalance
Keywords: Living donors; acute kidney injury; central venous pressure; Hemodynamic Monitoring; fluid therapy
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute kidney injury (AKI) is one of the most common complication after restricted fluid therapy for major surgery. The aim of this study is to evaluate the incidence of AKI as defined by Kidney Disease Improving Global Outcomes (KDIGO) criteria in living liver donor hepatectomy in which applied intraoperative protocolized fluid restriction targeting a low central venous pressure (CVP) level and high pulse pressure variation (PPV) / systolic pressure variation (SPV).

DETAILED DESCRIPTION:
Operative blood loss and need for transfusion are risk factors associated with mortality after partial hepatectomy. The low central venous pressure (CVP) anesthetic technique has been strongly advocated to minimize hepatic venous bleeding during hepatectomy. Low CVP technique for living donor hepatectomy may not be advantageous regarding the safety of healthy living donors. Safer, simpler, and more useful fluid management methods are, therefore, required to reduce blood loss and subsequent morbidity during living donor hepatectomy. Pulse pressure variation (PPV) and systolic pressure variation (SPV) are the dynamic parameters of hemodynamic used to access the volume status and fluid responsiveness in mechanically ventilated patients.

Based only on the serum creatinine increase, AKI occurs in 5-15% of hepatectomy patients.In this study, we aimed to evaluate the incidence of AKI based on the change of serum creatinine levels in living liver donor hepatectomy regarding intraoperative fluid restriction targeting low CVP levels and high PPV and SPV depending on our protocolized fluid management.

130 living liver donors were admitted for a retrospective observational study. The low central venous pressure (<5 mmHg) and high pulse pressure variation (PPV<20%) / systolic pressure variation (SPV<15%) were applied to reduce intraoperative blood loss as fluid management until the end of the hepatic parenchymal division. AKI was defined using the KDIGO criteria according to the serum creatinine. The SPSS 11.5 program was used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent living liver donor hepatectomy

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients who underwent living liver donor hepatectomy
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury in living donor patients | one week
  Kidney Disease Improving Global Outcomes (KDIGO) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Süheyla Karadağ Erkoç, Principal Investigator — Ankara University
Locations (1):
- Süheyla Karadağ Erkoç, Ankara, Turkey (Türkiye)